CLINICAL TRIAL: NCT03253887
Title: Effectiveness of Ethanol-Lock Therapy for the Prevention of Non-Tunneled Catheter-Related Bloodstream Infection in Pediatric Patients: A Randomised Controlled Trial
Brief Title: Ethanol-lock Therapy for the Prevention of Non-tunneled Catheter-related Infection in Pediatric Patients
Acronym: E-LockPed
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Collaborators: Bellisa Caldas Lopes (Unknown); Thuanne Beatriz Silva Tenório (Unknown); Rodrigo Melo Gallindo (Unknown); Paulo Sérgio Gomes Nogueira Borges (Unknown); Lara Barreto Machado (Unknown)
Responsible Party: Principal Investigator, Flavia orange, PhD, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 55008116.8.0000.5201
Record Dates: First submitted 2017-03-28; First posted 2017-08-18 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Infection, Catheter-Related; Central Line-associated Bloodstream Infection (CLABSI); Pediatric
Keywords: Central Venous Catheters; Child; ethanol therapy; CLABSI
MeSH Terms: conditions — Catheter-Related Infections | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: It's a randomized controlled clinical trial.
Who Masked: Outcomes Assessor
Masking Description: Following inclusion, the patients were randomized into two groups, the ethanol-lock group and the control group, using allocation concealment with a list of random numbers generated using the Random Allocation Software
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ethanol-lock therapy (ELT) Group (Experimental): This group received daily alcohol 70% (ethanol-lock) with intraluminal alcoholization of both lumens of the central venous catheters
  Interventions: Drug: Ethanol-lock
- Control Group (No Intervention): This group did not receive the ethanol-lock, being only followed daily and treated according to the standard protocol in operation at this healthcare unit.

INTERVENTIONS:
Drug: Ethanol-lock — This group received daily alcohol 70% (ethanol-lock) received intraluminal ethanol at a volume sufficient to fill the catheter lumen, ranged from 0.1 to 0.3 ml, with the volume being previously established. ELT was maintained for two full hours in each catheter lumen, with the lumen remaining locked during this period. The same procedure was then carried out with the other lumen. Prior to and following ELT, flushing was performed using 5-10 ml of 0.9% saline solution.
  Other Names: Ethanol 70%; Alcohol 70%
  Arms: Ethanol-lock therapy (ELT) Group

SUMMARY:
Central venous catheter (CVC) infection is a common complication in pediatric patients, resulting in prolonged length of stay in hospital, requiring antibiotics, invasive procedures and increase morbidity and mortality. Given the repercussion of this complication, measures that minimize its should be stimulated. The purpose of this study is to evaluate the effects of intraluminal alcoholization (ethanol lock therapy) on prevention of infection of short-term central venous catheters in pediatric patients.

DETAILED DESCRIPTION:
The patients was divided into two groups, where one received alcoholization (ethanol lock therapy group) and the other not (control group). The variables evaluated were: CLABSI, etiological agents, adverse events and the mechanical effects of ethanol on the catheter (breakage and obstruction). To determine the association between the independent variable and the dependent variables, the chi-square test of association (Pearson) and Fisher's exact test were used. The Risk Ratio (RR) was calculated as a relative risk measure, with its 95% confidence interval (95% CI). The significance level of 5% was adopted. The sample size calculation was performed in the OpenEpi software version 2.3.1. And a long-term catheter clinical trial was used to calculate the sample size, which demonstrated a 9% central venous catheter infection frequency in the ethanol group and 37% in the control group, so that the sample size was 80 patients (40 in each group), considering a power of 80%, an alpha error of 5% and 10% of post-randomization losses.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric surgery patients;
* Weight: 2 Kg or more;
* Using non-tunneled double-lumen polyurethane central venous catheter;
* CVC inserted at operation room, Pediatric Intensive Care Unit (PICU) or Neonatal Intensive Care Unit (NICU);
* CVC adequately positioned (checked by radioscopy ou radiography);
* CVC implanted within a maximum of 24 hours.

Exclusion Criteria:

* Patients whose catheters had been inserted under emergency situations;
* Patients in a critical condition (those requiring continuous fluid/drug infusion through both lumens);
* Patients with a history of hypersensitivity or allergic reactions to ethanol were excluded from the study.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Number of central line associated bloodstream infection (CLABSI) episodes in each group and compare them | Period from 48 hours after catheter insertion to 24 hours after catheter removal
  Measure of Central line associated bloodstream infection (CLABSI) rate per 1000 catheter-days compared between the groups, according to CDC's National Healthcare Safety Network (CDC/NHSN) 2015 definitions.

SECONDARY OUTCOMES:
main etiological agents involved in central line associated bloodstream infection (CLABSI) events | Considering that blood specimens were collected 48 hours after catheter insertion and up to 24 hours after catheter removal, from July 2016 to April 2017.
  The organisms responsable for each CLABSI event: gram negatives, gram positives or fungus. Identified by one or more blood specimens by a culture or non-culture based microbiologic testing method and the organism(s) identified in blood is not related to an infection at another site
Incidence of Treatment-Emergent Adverse Events | During the use of ethanol-lock therapy
  Number of episodes of adverse events (dizziness, headache, dyspnea, chest pain, alcohol taste, facial flushing, nausea, vomiting, pruritus, sneezing, slurred speech, irritability)
Incidence of mechanical effects of ethanol-lock on the catheter (catheter breakage and obstruction) | During the use of ethanol-lock therapy
  Evaluate mechanical effects of ethanol-lock on the catheter, by the number of participants with catheter breakage or catheter obstruction in each group

CONTACTS AND LOCATIONS:
Overall Officials: Bellisa C Lopes, Master, Principal Investigator — Instituto de Medicina Integral Prof Fernando Figueira
Locations (1):
- Instituto de Medicina Integral Prof Fernando Figueira, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flynn PM. Diagnosis and management of central venous catheter-related bloodstream infections in pediatric patients. Pediatr Infect Dis J. 2009 Nov;28(11):1016-7. doi: 10.1097/INF.0b013e3181bf7bfc. No abstract available. PMID 19859018
- [Background] Ullman AJ, Cooke ML, Mitchell M, Lin F, New K, Long DA, Mihala G, Rickard CM. Dressings and securement devices for central venous catheters (CVC). Cochrane Database Syst Rev. 2015 Sep 10;2015(9):CD010367. doi: 10.1002/14651858.CD010367.pub2. PMID 26358142
- [Background] Rosado V, Romanelli RM, Camargos PA. Risk factors and preventive measures for catheter-related bloodstream infections. J Pediatr (Rio J). 2011 Nov-Dec;87(6):469-77. doi: 10.2223/JPED.2134. PMID 22170387
- [Background] Subha Rao SD, Joseph MP, Lavi R, Macaden R. Infections related to vascular catheters in a pediatric intensive care unit. Indian Pediatr. 2005 Jul;42(7):667-72. PMID 16085967
- [Background] Cruzeiro PC, Camargos PA, Miranda ME. Central venous catheter placement in children: a prospective study of complications in a Brazilian public hospital. Pediatr Surg Int. 2006 Jun;22(6):536-40. doi: 10.1007/s00383-006-1671-2. Epub 2006 May 5. PMID 16736225
- [Background] Huang EY, Chen C, Abdullah F, Aspelund G, Barnhart DC, Calkins CM, Cowles RA, Downard CD, Goldin AB, Lee SL, St Peter SD, Arca MJ; 2011 American Pediatric Surgical Association Outcomes and Clinical Trials Committee. Strategies for the prevention of central venous catheter infections: an American Pediatric Surgical Association Outcomes and Clinical Trials Committee systematic review. J Pediatr Surg. 2011 Oct;46(10):2000-11. doi: 10.1016/j.jpedsurg.2011.06.017. PMID 22008341
- [Background] Webster J, Gillies D, O'Riordan E, Sherriff KL, Rickard CM. WITHDRAWN: Gauze and tape and transparent polyurethane dressings for central venous catheters. Cochrane Database Syst Rev. 2016 May 4;2016(5):CD003827. doi: 10.1002/14651858.CD003827.pub3. PMID 27144903
- [Background] Costello JM, Morrow DF, Graham DA, Potter-Bynoe G, Sandora TJ, Laussen PC. Systematic intervention to reduce central line-associated bloodstream infection rates in a pediatric cardiac intensive care unit. Pediatrics. 2008 May;121(5):915-23. doi: 10.1542/peds.2007-1577. PMID 18450894
- [Background] Wolf J, Shenep JL, Clifford V, Curtis N, Flynn PM. Ethanol lock therapy in pediatric hematology and oncology. Pediatr Blood Cancer. 2013 Jan;60(1):18-25. doi: 10.1002/pbc.24249. Epub 2012 Aug 21. PMID 22911535
- [Background] Shenep LE, Shenep MA, Cheatham W, Hoffman JM, Hale A, Williams BF, Perkins R, Hewitt CB, Hayden RT, Shenep JL. Efficacy of intravascular catheter lock solutions containing preservatives in the prevention of microbial colonization. J Hosp Infect. 2011 Dec;79(4):317-22. doi: 10.1016/j.jhin.2011.07.010. Epub 2011 Sep 25. PMID 21945067
- [Background] Wales PW, Kosar C, Carricato M, de Silva N, Lang K, Avitzur Y. Ethanol lock therapy to reduce the incidence of catheter-related bloodstream infections in home parenteral nutrition patients with intestinal failure: preliminary experience. J Pediatr Surg. 2011 May;46(5):951-6. doi: 10.1016/j.jpedsurg.2011.02.036. PMID 21616259
- [Background] Sanders J, Pithie A, Ganly P, Surgenor L, Wilson R, Merriman E, Loudon G, Judkins R, Chambers S. A prospective double-blind randomized trial comparing intraluminal ethanol with heparinized saline for the prevention of catheter-associated bloodstream infection in immunosuppressed haematology patients. J Antimicrob Chemother. 2008 Oct;62(4):809-15. doi: 10.1093/jac/dkn284. Epub 2008 Jul 11. PMID 18621987
- [Background] Chambers ST, Peddie B, Pithie A. Ethanol disinfection of plastic-adherent micro-organisms. J Hosp Infect. 2006 Jun;63(2):193-6. doi: 10.1016/j.jhin.2006.01.009. Epub 2006 Apr 4. PMID 16600429
- [Background] Abu-El-Haija M, Schultz J, Rahhal RM. Effects of 70% ethanol locks on rates of central line infection, thrombosis, breakage, and replacement in pediatric intestinal failure. J Pediatr Gastroenterol Nutr. 2014 Jun;58(6):703-8. doi: 10.1097/MPG.0000000000000354. PMID 24590214
- [Background] Crnich CJ, Halfmann JA, Crone WC, Maki DG. The effects of prolonged ethanol exposure on the mechanical properties of polyurethane and silicone catheters used for intravascular access. Infect Control Hosp Epidemiol. 2005 Aug;26(8):708-14. doi: 10.1086/502607. PMID 16156328
- [Background] Opilla MT, Kirby DF, Edmond MB. Use of ethanol lock therapy to reduce the incidence of catheter-related bloodstream infections in home parenteral nutrition patients. JPEN J Parenter Enteral Nutr. 2007 Jul-Aug;31(4):302-5. doi: 10.1177/0148607107031004302. PMID 17595439
- [Background] Chhim RF, Crill CM, Collier HK, Arnold SR, Pourcyrous M, Meibohm B, Christensen M. Ethanol lock therapy: a pilot infusion study in infants. Ann Pharmacother. 2015 Apr;49(4):431-6. doi: 10.1177/1060028015569881. Epub 2015 Jan 28. PMID 25632063
- [Background] Upadhyayula S, Kambalapalli M, Harrison CJ. Safety of anti-infective agents for skin preparation in premature infants. Arch Dis Child. 2007 Jul;92(7):646-7. doi: 10.1136/adc.2007.117002. No abstract available. PMID 17588981
- [Background] Mermel LA, Alang N. Adverse effects associated with ethanol catheter lock solutions: a systematic review. J Antimicrob Chemother. 2014 Oct;69(10):2611-9. doi: 10.1093/jac/dku182. Epub 2014 Jun 2. PMID 24891431
- [Background] Sharma V, Sharma A, Kumar V, Aggarwal S. Disulfiram-like reaction with ornidazole. J Postgrad Med. 2009 Oct-Dec;55(4):292-3. doi: 10.4103/0022-3859.58940. PMID 20083883
- [Background] Karamanakos PN, Pappas P, Boumba VA, Thomas C, Malamas M, Vougiouklakis T, Marselos M. Pharmaceutical agents known to produce disulfiram-like reaction: effects on hepatic ethanol metabolism and brain monoamines. Int J Toxicol. 2007 Sep-Oct;26(5):423-32. doi: 10.1080/10915810701583010. PMID 17963129
- Available data/document: Study Protocol — https://www.cdc.gov/nhsn/pdfs/pscmanual/4psc_clabscurrent.pdf — Bloodstream Infection Event (Central Line-Associated Bloodstream Infection and non-central line-associated Bloodstream Infection)
- Available data/document: Study Protocol — https://www.cdc.gov/nhsn/pdfs/pscmanual/17pscnosinfdef_current.pdf — CDC/NHSN Surveillance Definitions for Specific Types of Infections